CLINICAL TRIAL: NCT06450509
Title: Babble Boot Camp for Infants With Down Syndrome: Improving Speech and Language Outcomes Via a Proactive, Parent-led Intervention
Brief Title: Proactive Speech and Language Intervention for Infants With Down Syndrome
Acronym: BBC-DS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: American Speech-Language-Hearing Foundation (Other)
Responsible Party: Principal Investigator, Beate Peter, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00018407
Record Dates: First submitted 2024-02-29; First posted 2024-06-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-08

CONDITIONS: Down Syndrome
Keywords: Speech development; Language development; Linguistic environment; Parental stress; Babble complexity
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Participating infants and their parents will be randomized into two different treatment modalities, either weekly individualized intervention sessions or monthly group sessions. Both groups will receive the intervention for a duration of 10 months. Note that in each family, the infant and both caregivers, where available, will be enrolled. In each treatment arm, there will be 10 infants and up to 20 caregivers, for a total of 20 infants and up to 40 caregivers.
Who Masked: Outcomes Assessor
Masking Description: Individuals who analyze the audio recordings and score the questionnaires will not know the group assignments of the families.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individual intervention (Experimental): Individual families will meet weekly with a pediatric speech-language pathologist for approximately 20 minutes. The speech-language pathologist will coach parents in strategies designed to boost speech and language skills, individually tailored to the child's current skillset.
  Interventions: Behavioral: Babble Boot Camp
- Group intervention (Active Comparator): Caregivers will meet in monthly 1-hour group sessions with a pediatric speech-language pathologist. The speech-language pathologist will describe strategies that families can use at home to boost their child's speech and language skills.
  Interventions: Behavioral: Babble Boot Camp

INTERVENTIONS:
Behavioral: Babble Boot Camp — Caregivers are coached by a pediatric speech-language pathologist to implement activities and routines into their daily home lives with the intent to foster and boost their child's precursor and earliest speech and language skills. The intervention will be conducted entirely via telehealth.

SUMMARY:
Children with Down syndrome (DS) face life-long struggles with verbal communication. Babble and speech sound development is delayed, and speech can be difficult to understand. Words emerge late, at 21 months on average, compared to 12 months for typical peers, and vocabulary and grammar can remain limited throughout adulthood. Because DS is diagnosed at or even before birth, these difficulties are predictable; yet despite this prognostic knowledge, systematic and sustained proactive interventions have not yet been developed: Most children with DS are not assessed and treated for speech and language delays until age 2 to 4 years. This presents an untapped opportunity space to conduct a clinical trial of a proactive intervention in earliest infancy with the goal of building resilience against the anticipated difficulties. The intervention trialed here is a modified version of Babble Boot Camp (BBC), a proactive speech and language intervention originally developed for young infants with classic galactosemia (CG) (NIH 5R01HD098253). CG is a metabolic disease that, similar to DS, is diagnosed at birth and poses risks for severe speech and language delays. BBC is implemented by a speech-language pathologist who, via telehealth, trains parents to incorporate skill-building activities and routines into their daily lives at home. For the present study, 20 children with DS age birth to 12 months will be recruited and randomized into two treatment arms. One group will receive weekly individualized parent sessions and close monitoring of the child's progress. The second group will receive the same content but at a lower intensity and dosage, via monthly parent group meetings. Both groups will receive their intervention for 10 months. Specific aims are to quantify benefits for babble, speech production, and receptive and expressive language and to investigate associations between conversational dynamics in child-adult interactions and the children's speech and language. Outcomes in speech and language skills will show relative feasibility and benefits for each of these treatment modalities and motivate a larger clinical trial, with the ultimate goal of changing the way infants with DS receive support in their speech and language development, from a deficit-based, remedial model to a proactive one.

DETAILED DESCRIPTION:
Children with Down syndrome (DS) face life-long struggles with verbal communication. Babble and speech sound development is delayed, and speech can be difficult to understand. Words emerge late, at 21 months on average, compared to 12 months for typical peers, and vocabulary and grammar can remain limited throughout adulthood. Because DS is diagnosed at or even before birth, these difficulties are predictable; yet despite this prognostic knowledge, systematic and sustained proactive interventions have not yet been developed: Most children with DS are not assessed and treated for speech and language delays until age 2 to 4 years. This presents an untapped opportunity to conduct a clinical trial of a proactive intervention in earliest infancy with the goal of building resilience against the anticipated difficulties. The intervention trialed here is a modified version of Babble Boot Camp (BBC), a proactive speech and language intervention originally developed for young infants with classic galactosemia (CG) (NIH 5R01HD098253). CG is a metabolic disease that, similar to DS, is diagnosed at birth and poses risks for severe speech and language delays. BBC is implemented by a speech-language pathologist who, via telehealth, trains caregivers to incorporate skill-building activities and routines into their daily lives at home. For the present study, 20 children with DS age birth to 12 months will be recruited and randomized into one of two treatment arms. One group will receive weekly individualized caregiver sessions and close monitoring of the child's progress. The second group will receive the same content but at a lower intensity and dosage, via monthly caregiver group meetings. Both groups will receive their intervention for 10 months. At the beginning and end of the intervention, a set of data will be collected: At the beginning of the interventions, caregivers will be asked to complete an intake questionnaire with demographic information and information about the child's birth history, health history, and any services currently accessed. At the end of the intervention, caregivers will provide updates to this questionnaire and also a satisfaction survey. At pre and post, caregivers will provide three daylong audio recordings that will be analyzed for child utterance rates and conversational turns. For children age 6 months and up. these recordings will also be queried for segments with greatest numbers of child utterances, and these will be transcribed into International Phonetic Alphabet to obtain an objective measure of babble complexity, using the Mean Babbling Level, and, if sufficient numbers of meaningful utterances are found, an objective measure of word complexity using the Syllable Structure Level. At pre and post, questionnaires will be collected to appraise the children's general development and communication competence, using the Vineland Adaptive Behavior Scales 3. More detailed measures of early language skills, such as receptive and expressive vocabulary, will be obtained with the MacArthur-Bates Communicative Development Inventories -3. Age at emergence of first words will be recorded as a personal milestone for each child. Regarding parental well-being, the Parenting Stress Index 4 Short Form will be collected to obtain measures of stress originating in the parents themselves, in parent-child interactions, and in difficult child behaviors. This questionnaire also contains an estimate of whether or not parents are under-reporting their own personal stress. Specific aims are to quantify 1) benefits of each of the two interventions for babble and early speech sound production, 2) benefits of each of the two interventions for receptive and expressive language skills, and 3) associations between caregiver-child conversational dynamics during the intervention and child speech and language skill after the intervention. Outcomes in speech and language skills will show relative feasibility and benefits for each of these treatment modalities on children's speech and language development as well as parental well-being, and they will motivate a larger clinical trial, with the ultimate goal of changing the way infants with DS receive support in their speech and language development, from a deficit-based, remedial model to a proactive one.

ELIGIBILITY:
Inclusion Criteria:

* Full trisomy 21
* English is the main language spoken in the home

Exclusion Criteria:

* Partial or mosaic trisomy 21
* Any additional condition that could confound the findings
* Awaiting heart surgery
* Born prematurely before 34 weeks gestation

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Linguistic environment | Collected at the beginning of the intervention (baseline) and again at the end of the intervention (10 months later)
  Families will provide a set of three day-long audio recordings. Using the day-long audio recordings, the investigators will obtain adult word counts, child utterance counts, and conversational turn rates.
Child utterance complexity | Collected at the beginning of the intervention (baseline) and again at the end of the intervention (10 months later)
  Child utterance complexity will be based on the six day-long audio recordings that will be provided by the families in sets of three each. For children age 6 months and up, the investigators will mine the day-long audio recordings for those 5-minute segments with the highest numbers of child utterances. These utterances will be transcribed into the International Phonetic Alphabet. The utterances will be scored for phonetic complexity based on the consonant and vowel content. For babbled utterances, the investigators will compute the Mean Babbling Level (scores range from 1 to 3), and for meaningful utterances, the investigators will compute the Syllable Structure Level (scores range from 1 to 4). For both of these measures, higher scores reflect greater utterance complexity. Child utterance complexity will be based on the six day-long audio recordings that will be provided by the families in sets of three each at the beginning (baseline) and end (10 months later) of the intervention.
MacArthur-Bates Communicative Inventories 3: Comprehensive Parent | Collected at the beginning of the intervention (baseline) and again at the end of the intervention (10 months later)
  In this checklist-based questionnaires, caregivers provide information about their child's language skills, for instance how many words the child understands and how many words the child produces. Point scores are converted into percentiles, where higher numbers reflect better outcomes.
Vineland Adaptive Behavior Scales 3: Comprehensive Parent/Caregiver Form | Collected at the beginning of the intervention (baseline) and again at the end of the intervention (10 months later)
  Parents complete this questionnaire. Areas included in it are Communication, Daily Living Skills, Socialization, and Motor Skills. Point scores from the questionnaire are converted into standard scores and percentiles, where higher numbers reflect better outcomes.
Age at first words | This milestone may occur at any point through the 10 months of intervention, or not at all.
  For each child, the age at which she/he started to produce words is recorded.

SECONDARY OUTCOMES:
Consonant and vowel inventory | Collected at the beginning of the intervention (baseline) and again at the end of the intervention (10 months later)
  From the phonetic transcriptions of the day-long audio recordings, an inventory of consonant and vowel sounds will be made.
Parenting Stress Index 4 Short Form | Collected at the beginning of the intervention (baseline) and again at the end of the intervention (10 months later)
  In three blocks of 12 questions each, parents report on their own personal stress, stress derived from stressful interactions with the child, and stress derived from the child's difficult behaviors. Raw scores are converted into percentiles. Higher percentiles indicate higher levels of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Beate Peter, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified information will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be shared starting in February 2025 for a period of 5 years.
Access Criteria: Qualified researchers must contact the PI to request access to the data.

REFERENCES:
- [Background] Potter NL, VanDam M, Bruce L, Davis J, Eng L, Finestack L, Heinlen V, Scherer N, Schrock C, Seltzer R, Stoel-Gammon C, Thompson L, Peter B. Virtual Post-Intervention Speech and Language Assessment of Toddler and Preschool Participants in Babble Boot Camp. J Speech Lang Hear Res. 2024 Sep 26;67(9S):3327-3339. doi: 10.1044/2023_JSLHR-22-00687. Epub 2023 May 26. PMID 37235746
- [Background] Peter B, Bruce L, Finestack L, Dinu V, Wilson M, Klein-Seetharaman J, Lewis CR, Braden BB, Tang YY, Scherer N, VanDam M, Potter N. Precision Medicine as a New Frontier in Speech-Language Pathology: How Applying Insights From Behavior Genomics Can Improve Outcomes in Communication Disorders. Am J Speech Lang Pathol. 2023 Jul 10;32(4):1397-1412. doi: 10.1044/2023_AJSLP-22-00205. Epub 2023 May 5. PMID 37146603
- [Background] Finestack LH, Potter N, VanDam M, Davis J, Bruce L, Scherer N, Eng L, Peter B. Feasibility of a Proactive Parent-Implemented Communication Intervention Delivered via Telepractice for Children With Classic Galactosemia. Am J Speech Lang Pathol. 2022 Nov 16;31(6):2527-2538. doi: 10.1044/2022_AJSLP-22-00107. Epub 2022 Oct 14. PMID 36251874
- [Background] Peter B, Davis J, Finestack L, Stoel-Gammon C, VanDam M, Bruce L, Kim Y, Eng L, Cotter S, Landis E, Beames S, Scherer N, Knerr I, Williams D, Schrock C, Potter N. Translating principles of precision medicine into speech-language pathology: Clinical trial of a proactive speech and language intervention for infants with classic galactosemia. HGG Adv. 2022 May 20;3(3):100119. doi: 10.1016/j.xhgg.2022.100119. eCollection 2022 Jul 14. PMID 35677809
- [Background] Peter B, Davis J, Cotter S, Belter A, Williams E, Stumpf M, Bruce L, Eng L, Kim Y, Finestack L, Stoel-Gammon C, Williams D, Scherer N, VanDam M, Potter N. Toward Preventing Speech and Language Disorders of Known Genetic Origin: First Post-Intervention Results of Babble Boot Camp in Children With Classic Galactosemia. Am J Speech Lang Pathol. 2021 Nov 4;30(6):2616-2634. doi: 10.1044/2021_AJSLP-21-00098. Epub 2021 Oct 19. PMID 34665663
- [Background] Peter B, Potter N, Davis J, Donenfeld-Peled I, Finestack L, Stoel-Gammon C, Lien K, Bruce L, Vose C, Eng L, Yokoyama H, Olds D, VanDam M. Toward a paradigm shift from deficit-based to proactive speech and language treatment: Randomized pilot trial of the Babble Boot Camp in infants with classic galactosemia. F1000Res. 2019 Mar 11;8:271. doi: 10.12688/f1000research.18062.5. eCollection 2019. PMID 32566130